CLINICAL TRIAL: NCT07223489
Title: Understanding the Diagnostic Pathway and Treatment Experience of Patients With Spinal Muscular Atrophy (SMA)
Brief Title: Diagnostic Journey, Patient Experience, and Disparities in the Treatment of Spinal Muscular Atrophy (SMA) in the MedStar Health System
Acronym: SMA
Status: Recruiting | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Principal Investigator, Nicholas Streicher, Physician, Medstar Health Research Institute
Other Study IDs: ML46436
Record Dates: First submitted 2025-10-29; First posted 2025-10-31 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Spinal Muscular Atrophy (SMA)
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Telephone Interview — Telephone interviews to gather qualitative data on SMA patients' diagnostic journey, access to treatment and barriers encountered, understanding of their disease, and quality of life measures

SUMMARY:
Evaluate the diagnostic journey, patient experience, and disparities in the treatment of Spinal Muscular Atrophy (SMA) in the MedStar Health System.

DETAILED DESCRIPTION:
Spinal Muscular Atrophy (SMA) is a genetic neuromuscular disorder caused by mutations in the SMN1 gene, leading to degeneration of motor neurons and progressive muscle weakness. While disease-modifying therapies such as nusinersen (Spinraza), onasemnogene abeparvovec-xioi (Zolgensma), and risdiplam (Evrysdi) have significantly improved outcomes for individuals with SMA, access to these treatments remains inconsistent-especially among adults. Many adults with SMA remain untreated or experience long delays in diagnosis and initiation of therapy, reflecting potential gaps in awareness, care coordination, and health equity.

This observational, two-phase study will evaluate the diagnostic pathways and treatment experiences of SMA patients receiving care within the MedStar Health System.

Phase 1 (Retrospective Chart Review): Medical records will be reviewed to characterize diagnostic timelines, genetic confirmation, treatment history, and demographic variables. This phase will identify eligible participants for qualitative interviews and describe patterns of treatment uptake and care access.

Phase 2 (Qualitative Interviews): Eligible patients aged 18 years or older will be invited to participate in one-time telephone interviews lasting approximately 60 minutes. Interviews will explore patients' diagnostic experiences, understanding of their condition, access to therapies, barriers encountered, and perceived quality of care.

The study will enroll up to 200 participants, beginning with the Georgetown Neurology clinic and expanding across the MedStar Health network. Participation involves minimal risk. The primary risks are potential discomfort in discussing personal health experiences and loss of confidentiality, which will be minimized through secure data handling procedures, staff training, and voluntary participation.

Results will inform strategies to improve SMA diagnosis and care pathways, particularly among underserved populations. Findings may also support health system initiatives to reduce disparities in access to specialized neuromuscular care.

ELIGIBILITY:
Inclusion Criteria:

* SMA diagnosis, age greater than or equal to 18 years

Exclusion Criteria:

* Deceased

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SMA patients within the MedStar Health Network
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-10-10 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of SMA patients not receiving disease-modifying therapy and categorical causes for non-treatment based on structured patient/caregiver survey responses | 2020-2025
  The primary outcome assesses the percentage of patients with a confirmed diagnosis of spinal muscular atrophy (SMA) who are not currently receiving an FDA-approved disease-modifying therapy (nusinersen, risdiplam, or onasemnogene abeparvovec). Data are collected through a structured telephone or in-person survey using the Lost to Follow-Up Interview Questionnaire, designed to identify categorical reasons for non-treatment. Categories include insurance or financial barriers, clinical contraindications, patient preference, adverse effects, loss to follow-up, or access limitations. The outcome will quantify the proportion of patients in each category to identify predominant causes of non-treatment and guide future outreach and care re-engagement strategies.
  Unit of Measure:
  Percentage of participants.

CONTACTS AND LOCATIONS:
Locations (1):
- MedStar Health Research Institute, Washinton, District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No